CLINICAL TRIAL: NCT00263679
Title: A Phase III, Double-blinded, Randomized, Multicenter, Clinical Study to Assess the Safety and Immunogenicity of GSK Biologicals' Tdap 0.3 mg Candidate Vaccine When Given as a Booster Dose to Healthy School Children and Adolescents (9-13 Years of Age), Previously Vaccinated With a 5th Consecutive Dose of Acellular Pertussis-containing Vaccine, in Studies APV-118 or APV-120
Brief Title: Assessment of GSK Biologicals' Tdap Candidate Vaccine Administered as a Booster (6th Dose) in Terms of Immunogenicity and Safety to Children and Adolescents Previously Vaccinated With Five Doses of an Acellular Pertussis-containing Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 100406/004
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Acellular Pertussis; Diphtheria; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: Prophylaxis: Diphtheria, tetanus and pertussis

SUMMARY:
The aims of this study are to evaluate the safety and immunogenicity of a booster dose of GSK Biological's candidate Tdap vaccine containing 0.3 mg Al when administered to healthy school children and adolescents (9-13 years of age) previously vaccinated with five consecutive doses of Pa-containing vaccine. The inclusion of hepatitis A vaccine (Havrix®) as a control vaccine enables this study to be conducted in a double-blinded in terms of immunogenicity and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

- Subjects previously enrolled and vaccinated in GSK Biologicals' studies APV-118 and APV-120 and who were 9 through 13 years of age

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the administration of study vaccines, or planned use during the study period.
* Chronic administration or planned administration of immunosuppressants or other immune modifying drugs within six months prior to study vaccination or planned administration during the study period
* Administration of immunoglobulins and/or blood products within 3 months prior to vaccination

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2003-11; Primary Completion 2004-05 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Safety after vaccination.

SECONDARY OUTCOMES:
Immunogenicity and safety after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Germany (10):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Limburg an der Lahn, Hesse
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Mertsola J et al. The immunogenicity and safety of repeated administration of dTpa booster in adolescents and young adults. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Mertsola J et al. The safety of repeated administration of Boostrix™, a reduced-antigen-content dTpa booster. Abstract presented at Excellence In Paediatrics (EIP). Florence, Italy, 3-6 December 2009.
- [Background] Mertsola J et al. The safety of repeated administration of reduced-antigen-content dTpa boosters. Abstract presented at WSPID- 6th World Congress. Buenos Aires, Argentina, 19-22 November 2009
- [Background] Zepp F, Knuf M, Habermehl P, Mannhardt-Laakmann W, Howe B, Friedland LR. Safety of reduced-antigen-content tetanus-diphtheria-acellular pertussis vaccine in adolescents as a sixth consecutive dose of acellular pertussis-containing vaccine. J Pediatr. 2006 Nov;149(5):603-610. doi: 10.1016/j.jpeds.2006.06.016. PMID 17095328
- [Background] Zepp F, Habermehl P, Knuf M, Mannhardt-Laakman W, Howe B, Friedland LR. Immunogenicity of reduced antigen content tetanus-diphtheria-acellular pertussis vaccine in adolescents as a sixth consecutive dose of acellular pertussis-containing vaccine. Vaccine. 2007 Jul 20;25(29):5248-52. doi: 10.1016/j.vaccine.2007.05.012. Epub 2007 Jun 4. PMID 17583395
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100406/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register